CLINICAL TRIAL: NCT05473195
Title: A Phase 2 Trial to Evaluate the EBA, Safety and Tolerability of Ethionamide Alone and in Combination With BVL-GSK098 Administered Orally to Adults With Newly Diagnosed, Rifampicin- and Isoniazid-Susceptible Pulmonary Tuberculosis
Brief Title: A Phase 2 Trial to Evaluate the EBA, Safety and Tolerability of Eto Alone and in Combination With BVL-GSK098
Acronym: BETO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TASK Applied Science (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASK-010-BETO
Record Dates: First submitted 2022-07-12; First posted 2022-07-25 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Rifampicin- and Isoniazid-Susceptible Pulmonary Tuberculosis (TB)
MeSH Terms: interventions — Ethionamide; Isoniazid

STUDY DESIGN:
Intervention Model Description: A single-centre, open-label, clinical trial in two stages. All treatments will be administered orally (PO) on days 1-7.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm 1 (Experimental): BVL-GSK098 9 mg once daily (OD) plus ethionamide 250 mg OD (b9Eto250)
  Interventions: Drug: BVL-GSK098 9mg; Drug: Ethionamide 250mg
- Arm 2 (Active Comparator): Isoniazid 300 mg po OD (INH)
  Interventions: Drug: Isoniazid 300 MG
- Arm 3 (Experimental): BVL-GSK098 27 mg OD plus ethionamide 125 mg po OD (b27Eto125)
  Interventions: Drug: BVL-GSK098 9mg; Drug: Ethionamide 250mg
- Arm 4 (Experimental): BVL-GSK098 27 mg OD plus ethionamide 250 mg po OD (b27Eto250)
  Interventions: Drug: BVL-GSK098 9mg; Drug: Ethionamide 250 mg
- Arm 5 (Experimental): BVL-GSK098 27 mg OD plus ethionamide 500 mg po OD (b27Eto500)
  Interventions: Drug: Ethionamide 250mg
- Arm 6 (Experimental): Ethionamide 250 mg po OD (Eto250)
  Interventions: Drug: Ethionamide 250 mg
- Arm 7 (Experimental): Ethionamide 750 mg po given in a single or divided dose daily (Eto750)
  Interventions: Drug: Ethionamide 250mg

INTERVENTIONS:
Drug: BVL-GSK098 9mg — BVL-GSK098 9 mg once daily po OD plus ethionamide 250 mg po OD (b9Eto250) BVL-GSK098 27 mg OD plus ethionamide 125 mg po OD (b27Eto125 BVL-GSK098 27 mg OD plus ethionamide 250 mg po OD (b27Eto250) BVL-GSK098 27 mg OD plus ethionamide 500 mg po OD (b27Eto500)
  Other Names: Ethionamide 125 and 250mg
  Arms: Arm 1; Arm 3; Arm 4
Drug: Ethionamide 250mg — Ethionamide 250 mg po OD (Eto250)
  Arms: Arm 1; Arm 3; Arm 5; Arm 7
Drug: Ethionamide 250 mg — Ethionamide 750 mg po given in a single or divided dose (Eto750)
  Other Names: Ethionamide 250mg
  Arms: Arm 4; Arm 6
Drug: Isoniazid 300 MG — Isoniazid 300 mg po OD (INH)
  Arms: Arm 2

SUMMARY:
To evaluate the 7-day early bactericidal activity (EBA), pharmacokinetics (PK), safety and tolerability of ethionamide (Eto) with or without BVL-GSK098 in participants with rifampicin- and isoniazid-susceptible pulmonary TB.

DETAILED DESCRIPTION:
A single-centre, open-label, clinical trial in two stages. All treatments will be administered orally (PO) on days 1-7.

Stage 1 will recruit 15 participants into arm 1 who will receive Eto and a low dose BVL-GSK098 combination (bEto), including 3 participants from the control arm (arm 2). Participants will be randomized 5:1. This will be followed by a recruitment pause and an interim analysis to evaluate safety of the combination.

Stage 1:

Arm Regimen Participants

1. BVL-GSK098 9 mg once daily (OD) plus ethionamide 250 mg OD (b9Eto250) 15
2. Isoniazid 300 mg po OD (INH) 3 * BVL-GSK098 9 mg will be given 12-hourly on Day one (loading dose), then once daily on Day 2-7.

An interim safety analysis will be performed after all Stage 1 participants complete the end of treatment visit (Day 8). If the b9Eto250 arm meets the predefined safety criteria (Section 9), the study will proceed to Stage 2. Recruitment will then continue with the remaining arms randomized in a 4:5:5:5:5:5 ratio.

Stage 2:

Arm Regimen Participants 2 Isoniazid 300 mg po OD (INH) 12 3 BVL-GSK098 27 mg OD plus ethionamide 125 mg po OD (b27Eto125) 15 4 BVL-GSK098 27 mg OD plus ethionamide 250 mg po OD (b27Eto250) 15 5 BVL-GSK098 27 mg OD plus ethionamide 500 mg po OD (b27Eto500) 15 6 Ethionamide 250 mg po OD (Eto250) 15 7 Ethionamide 750 mg po given in a single or divided dose daily (Eto750) 15

* BVL-GSK098 27 mg will be given 12-hourly on Day one (loading dose), then once daily on Day 2-7. Ethionamide 750 mg given in divided doses Day 1-3, and OD Day 4-7.

Participants on INH will serve as control for the EBA quantitative mycobacteriology. The study will not be blinded but the mycobacteriology laboratory staff performing the endpoint assays will remain blinded until analysis of the EBA results.

ELIGIBILITY:
Inclusion Criteria:

- Participants are required to meet all the following criteria in order to be randomized.

1. Provide written, informed consent prior to all trial-related procedures.
2. Male or female, aged between 18 and 65 years, inclusive.
3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Newly diagnosed and untreated pulmonary TB.
5. Rifampicin- and isoniazid-susceptible pulmonary TB as determined by molecular testing (GeneXpert XDR or Genotype MTBDRplus for INH).
6. A chest X-ray taken during the screening period or up to 2 weeks before screening which, in the opinion of the investigator, is consistent with TB.
7. GeneXpert positive with a quantitative readout of medium or high.
8. Ability to produce an adequate volume of sputum as estimated from an overnight sputum collection sample (estimated 10 ml or more).
9. Be of non-childbearing potential or using effective methods of birth control.
10. For WOCBP, injectable or other contraceptive methods (per Appendix 1) need to be given prior to or during screening, and at least 2 days prior to first dose of IP.

    Exclusion Criteria:
    * Participants will be excluded from participation if they fulfil any of the following criteria.

    Medical History
11. Evidence of clinically significant conditions or findings, other than TB, that might compromise safety or the interpretation of trial endpoints, per discretion of the investigator.
12. History of epilepsy, seizures or other neuropsychiatric disorders that might compromise safety or the interpretation of trial endpoints, per discretion of the investigator
13. History of hypothyroidism
14. QTcF of >450 ms at baseline
15. Clinically significant evidence of extrathoracic TB, as judged by the investigator.
16. History of allergy to any of the trial IP as confirmed by the clinical judgement of the investigator.
17. Alcohol or drug abuse, that in the opinion of the investigator, is sufficient to compromise the safety or cooperation of the participant.
18. HIV positive AND:

    1. CD4 < 250cells/mm3
    2. OR, on ART in stage 1 only. Participants established on ART (2 NRTIs and dolutegravir) for more than 30 days at start of screening are eligible for participation in stage 2.

    NOTE: ART permitted in Stage 2 is limited to the following in line with local guidelines for 1st line ART:
    * NRTIs selected from: Emtricitabine, Lamivudine, Tenofovir
    * PLUS Dolutegravir

    As the drug-drug interaction potential of ART has not been fully investigated with the IP, NNRTIs (efavirenz, nevirapine) and other protease inhibitors will not be permitted in this study.
19. Female participant who is pregnant, breast-feeding, or planning to conceive a child within the anticipated period of trial participation. Male participant planning to conceive a child for at least 90 days, after the last dose of study intervention in the trial.

    Treatment History
20. Participation in other clinical studies with investigational agents within 8 weeks prior to screening.
21. Treatment received for this episode of TB with any drug active against M.tb (including but not limited to isoniazid, ethambutol, amikacin, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides).
22. Treatment with immunosuppressive medications such as TNF-alpha inhibitors within 2 weeks prior to screening, or systemic corticosteroids for more than 7 days within 2 weeks prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
EBA CFU | 7 days
  The EBA CFU(0-7) as determined by the predicted rate of change in log10CFU per ml sputum over the period day 0 to day 7 will be described using linear, bi-linear or non-linear functions using nonlinear mixed effects modelling as dictated by the data of log10CFU over time and relation to drug exposure.
  Predicted estimate of rates of change including uncertainties for the potential differences in treatment effects between the groups will be given and graphically illustrated.

SECONDARY OUTCOMES:
EBA TTP | 7 days
  The EBA TTP(0-7) as determined by the predicted rate of change in TTP over the period day 0 to day 7 will be described using linear, bi-linear or non-linear functions using nonlinear mixed effects modelling of TTP over time and relation to drug exposure.

OTHER OUTCOMES:
Adverse events | 7 days
  The incidence of the following events will be summarized by treatment group:
  * Incidence of treatment-emergent adverse events (TEAEs);
  * Incidence of TEAEs by Severity;
  * Incidence of drug related TEAEs;
  * Incidence of Serious TEAEs;
  * Incidence of TEAEs leading to early withdrawal;
  * Incidence of TEAEs leading to death.
  Descriptive summary statistics will be presented for other safety variables: laboratory parameters, physical examination, vital signs, concomitant medication.

CONTACTS AND LOCATIONS:
Overall Officials: Reinard McPherson, MBChB, Principal Investigator — TASK
Locations (1):
- TASK Clinical Research Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Plan not yet available
Supporting Information: Study Protocol
Time Frame: Immediately after publication.
Access Criteria: Not available yet